CLINICAL TRIAL: NCT00777985
Title: Cardiovascular Consequences of Obstructive Sleep Apnea (OSA): Role of Endothelin and Preventive Effects of Bosentan
Brief Title: Preventive Effects of Bosentan on the Systemic Cardiovascular Consequence of Sleep Apnea
Acronym: BOSAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0722; 2007-005333-11 (Registry Identifier: EudraCT number)
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea; Hypertension
Keywords: Cardiovascular system; Sleep; Endothelial function; Endothelin system
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — Bosentan; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bosentan
- 2 (Active Comparator)
  Interventions: Device: nasal continuous positive airway pressure (CPAP)

INTERVENTIONS:
Drug: bosentan — 62.5 mg b.i.d for 4 weeks
  Other Names: TRACLEER
  Arms: 1
Device: nasal continuous positive airway pressure (CPAP) — Daily application throughout sleep for 4 weeks
  Arms: 2

SUMMARY:
The study will compared the effects of bosentan, an endothelin receptor antagonist, and nasal continuous positive airway pressure (nCPAP), obstructive sleep apnea current reference treatment, on diastolic blood pressure in untreated mildly hypertensive sleep apnea patients.

The hypothesis is that blocking endothelin receptors with a drug will have the same systemic blood pressure lowering effect than nCPAP in sleep apnea patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented obstructive sleep apnea
* with untreated mild systemic hypertension

Exclusion Criteria:

* pregnancy or lactation
* daytime alveolar hypoventilation
* severe arterial hypertension (systolic pressure > 180 mmHg; diastolic pressure > 110 mmHg)
* treatment with anti-hypertensive drugs
* cardiovascular disorder other than mild hypertension
* severe daytime sleepiness (score on the EPWORTH sleepiness scale ≥15) or at-risk occupation
* contra-indication to nCPAP treatment
* known allergy to bosentan
* active treatment with a drug whose efficacy is reduced by cytochromes P450, 2C9, 3A4 and2C19 isoenzyme activation
* active treatment with a drug acting on systemic arterial blood pressure or endothelial function
* liver or kidney dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
24 hour mean diastolic blood pressure | before and after each treatment completion (4 weeks)

SECONDARY OUTCOMES:
Peripheral Arterial Tonometry measure | before and after each treatment completion (4 weeks)
mean 24 hour systemic systolic blood pressure | before and after each treatment completion (4 weeks)
mean 24 hour nocturnal blood pressure | before and after each treatment completion (4 weeks)
carotid Intima Media Thickness | before and after each treatment completion (4 weeks)
Circulating inflammation markers (RANTES, MCP-1, TNF-alpha, INF-gamma, IL-6, IL-10 and TGF-gamma | before and after each treatment completion (4 weeks)
Circulating Big ET1 and ET1 levels | before and after each treatment completion (4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine H Launois, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de Grenoble, Grenoble, France

REFERENCES:
- [Result] Joyeux-Faure M, Jullian-Desayes I, Pepin JL, Cracowski JL, Baguet JP, Tamisier R, Levy P, Godin-Ribuot D, Launois SH. Comparison of continuous positive airway pressure and bosentan effect in mildly hypertensive patients with obstructive sleep apnoea: A randomized controlled pilot study. Respirology. 2016 Apr;21(3):546-52. doi: 10.1111/resp.12713. Epub 2015 Dec 8. PMID 26643404